CLINICAL TRIAL: NCT05693636
Title: Clinical and Patient-reported Outcomes After Total Wrist Arthroplasty and Total Wrist Arthrodesis: A Prospective Cohort-study With 2-year Follow-up
Brief Title: Clinical and Patient-reported Outcomes After Total Wrist Arthroplasty and Total Wrist Arthrodesis
Status: Completed | Type: Observational
Sponsor: Region Skane (Other)
Responsible Party: Sponsor
Other Study IDs: 2015/121
Record Dates: First submitted 2022-12-28; First posted 2023-01-23 (Actual); Last update posted 2023-01-23 (Actual); Status verified 2022-12

CONDITIONS: Wrist Arthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Total Wrist Fusion: Patients with end-stage wrist arthritis treated with total wrist fusion.
- Total Wrist Arthroplasty: Patients with end-stage wrist arthritis treated with total wrist arthroplasty of the fourth generation
  Interventions: Procedure: Total wrist arthroplasty

INTERVENTIONS:
Procedure: Total wrist arthroplasty — Two different surgical interventions for treatment of end-stage arthritis are compared
  Other Names: Total wrist fusion
  Groups: Total Wrist Arthroplasty

SUMMARY:
The wrist is often considered to be the fundament of the hand. Patients with a destroyed wrist joint caused by osteoarthritis or rheumatoid arthritis may suffer from pain and functional disabilities with impaired life quality.

The traditional surgical solution for advanced wrist arthritis is a total wrist fusion (TWF). Although TWF creates a stable wrist with minimal pain, the prize is the joint motion. Total wrist arthroplasty (TWA) is a motion-preserving alternative, but has failed to achieve the widespread use of other joint replacement procedures. TWA is more costly and technically demanding than TWF, and also associated with more complications. In addition, there is no consensus regarding the functional benefit of a TWA compared to TWF since prospective, comparative studies are missing.

Aim: The purpose of this prospective cohort study was to compare functional outcome and activity limitations up to two years after surgery with TWA or TWF.

DETAILED DESCRIPTION:
Patients with advanced wrist arthritis engaging both the midcarpal- and radiocarpal joints may suffer from pain, decreased joint motion and reduced grip strength. The traditional surgical solution with TWF creates a stable wrist with decreased pain, but the prize is the loss of wrist motion. TWA may be a motion-preserving alternative, but is more technically demanding and is associated with more complications compared to TWF. In addition, the functional benefits of TWA over TWF are still unknown.

Aim: The purpose of this prospective cohort study was to compare functional outcome and activity limitations up to two years after surgery with TWA or TWF.

Methods: In this single-center prospective, longitudinal cohort-study, all patients treated with TWF or TWA due to end-stage wrist arthritis at one hand surgical department between March 1, 2015, through February 28, 2020, were enrolled.The treatment method was decided by the treating consultant in hand surgery, based on clinical evaluation of the patient and radiographic appearance of the wrist, in combination with the patients' own requests and prerequisites.

Assessments were performed at baseline, 3 months, 6 months, 12 months and 24 months after surgery with patient-reported outcome measures, range-of-motion, grip strength and radiographic evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Both radoiocarpal and mid carpal arthritis due to osteoarthritis, inflammatory arthritis (such as rheumatoid/psoriasis arthritis), Kienböck's disease

Exclusion Criteria:

* Wrist problems due to hypermobility or cerebral palsy
* Severe cognitive disorder and unable to fill in questionnaires

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients seeking at one hand surgical department with wrist end-stage arthritis and planned for surgery with TWF or TWA were invited to participate in this study. The indications for either a TWF or a TWA at our department are: 1) severe wrist pain and functional disabilities, and 2) radiological evidence of end-stage arthritis, where other options such as proximal row carpectomy or partial arthrodesis are ruled out, and/or 3) the patient had undergone previous surgical procedure/s such as wrist arthroscopy, proximal row carpectomy or partial arthrodesis, but with insufficient results.
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2015-03-01 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Patient-Rated Wrist Evaluation (PRWE) at 24 months | Up to 24 months
  The PRWE is a self-reported questionnaire that includes 15 questions, divided into two subscales assessing pain (5 items) and function (10 items, 6 concerning specific tasks and 4 the ability to perform daily activities) over the past week. The questions are scored on a 10-point ordered categorical scale, ranging from no pain or no difficulty (0 points), to worst pain or unable to do (10 points). The total score of the subscales pain (sum of 5 items) and function (sum of 10 items divided by 2) ranges from 0 to 50. The maximum total score of PRWE is 100 and represents the worst disability, whereas 0 represents no disability.

SECONDARY OUTCOMES:
Visual Analoge Scale (VAS) pain at rest and on load | Up to 24 months
  Patients are rating pain in their wrist at a Visual Analoge Scale, ranging from 0-100, ranging from 0 (no pain) to 100 (most severe pain).
Grip strength | Up to 24 months
  Grip strength were assessed with a dynamometer in both hands. Three trials were recorded for each hand.
Disability of the Hand, Shoulder and Arm (DASH) | Up to 24 months
  The DASH questionnaire is a self-reported outcome measure, scored from 0 (no disability) to 100 (severe disability) and evaluates the function in the entire upper extremity.

OTHER OUTCOMES:
Radiographic evaluation | Up to 24 months
  Standard wrist radiographs (posterior anterior and lateral views) are obtained to verify and classify the arthritis preoperatively and to evaluate union in TWF-patients and osteolysis/loosening in TWA-patients

IPD SHARING:
Plan to Share IPD: No